CLINICAL TRIAL: NCT03747471
Title: Effect of Conversation Map on Diabetes Management Self-efficacy and Diabetic Distress Among Type 2DM Patient in Pakistan: A Randomized Controlled Trial
Brief Title: Conversation Map and Diabetes in Pakistan
Acronym: DAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rubina Qasim (Other)
Responsible Party: Sponsor-Investigator, Rubina Qasim, Lecturer, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ruby1234
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus; Diabetes; Self Efficacy; Diabetes Mellitus, Type 2
Keywords: Diabetes; Type 2 Diabetes mellitus; Health Education; Conversation Map; Developing countries
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Intervention Model Description: This will be a 2 arms individual randomized controlled trial. Intervention arm will receive teaching from the nurses using diabetic conversation map with visual images and control arm will receive teaching from the nurses using the traditional diabetic counselling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Intervention: Diabetic Conversation Map x 4 Sessions
  Interventions: Behavioral: Diabetic Conversation Map
- Control Arm (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Diabetic Conversation Map — Diabetic Conversation Map education tools are a series of tools for facilitated group education 5-8that were developed by Healthy Interactions in collaboration with the International Diabetes Federation (IDF) and are sponsored by Lilly Diabetes.
  CM-based education guides people with diabetes through a process with the aim of helping them understand and internalize information about their disease and generate insightful conclusions, which may then result in improved self-management decisions and actions.
  Arms: Experimental Arm

SUMMARY:
Background Diabetes is recognized as an important cause of premature death and disability. Non-clinical interventions play an important role in the control of diabetes and the prevention of its associated complications. Traditional methods of educating diabetic patients to empower them for the control of their disease might not work in the developing world. However, the novel interactive and pictorial health education tool named Diabetes Conversation Map (DCM) might be effective for the improvement of diabetes management self-efficacy and distress among diabetic patients in lower middle income setting of Karachi, Pakistan.

Objective To assess the effectiveness of DCM as compared to routine care to improve the diabetes management self-efficacy (DMSE) and diabetic distress (DD) among type 2 diabetic patients (T2DM) visiting diabetic clinics of tertiary care hospitals in lower middle income setting of Karachi, Pakistan.

Methodology This will be a two arms randomized controlled trial, conducted in two tertiary care hospitals, Karachi. A sample of 120 T2DM patients of age 30 - 60 years with sub-optimal diabetes control will be screened through eligibility criteria and diabetes distress screening tool. Patients who fulfill the eligibility criteria and have diabetes distress will be randomized into intervention (n=60) and control group (n=60) using sealed envelopes. The intervention arm will receive four diabetic education sessions using the DCM in a group of 5-8 participants and each session will be at the interval of one (1) week, by the principal investigator. T2DM patients in the controlled arm will receive routine care. Data on DMSE and DD will also be measured 2-3 months post intervention after the completion of all education sessions. Descriptive statistics will be used for data analysis through SPSS version 20; whereas, application of Repeated Measures ANOVA will be carried out for inferential statistics.

DETAILED DESCRIPTION:
Like any other chronic disease, the control of diabetes is very essential. Non-clinical interventions such as life style modification, stress relief and healthy dietary habits have been proven to be effective against the control of diabetes and prevention of diabetes related complications. Traditionally, diabetic patients used to receive education related to their disease process, metabolic control, exercise and diabetic diet through didactic lectures, brochures, pamphlets, and face to face counseling. While these traditional methods are found to be effective in diabetes self-management in the western world due to better literacy rate, level of understanding and access to modern modes of communications. However, in the developing world these methods could not work because of several reasons including poor literacy. Among novel methods, Diabetes Conversation Maps are considered as useful tools for the educational empowerment of diabetic patients. These are interactive pictorial tools designed in such a way that it does not need formal education for common understanding. In developing countries like Pakistan, where the literacy rate is very less, these tools might prove to be effective for the control of diabetes and its associated complications. Diabetes conversation maps have been used and tested in several countries predominantly in the developed world. In the developing region, while it has shown some impact during the observational studies, literature generated from randomized control trials is still limited. Patients in the developing region has different level of education and environmental exposures such as access to internet and social media, they have different socio-demographic characteristics and hence might behave differently from their counterparts in the developed world. Therefore, there is a need of well-designed randomized controlled trial to evaluate the effectiveness of Diabetes Conversation Map versus routine diabetic care in DMSE and DD in a low middle income setting of Karachi, Pakistan.

Research Question Is effectiveness of DCM as an educational tool same as routing care for improving the DMSE and DD in patients with T2DM visiting diabetic clinic of a tertiary care hospital in Karachi, Pakistan? 1.2 Significance of study: This study is a pioneer effort for generating new knowledge about the use of Diabetes Conversation Map. Findings of this study will be helpful for the nursing leadership and organizational leadership for use of Diabetes Conversation Map for managing the risks factors / complications of the DM. Also, it is cost effective intervention to be implemented by the health professionals, resulting in saving patients from managing DM, its complications, money and time. Moreover, findings of this study will be available for Pakistan Nursing Council (PNC) and Pakistan Medical and Dental Council (PMDC), for inculcating it into the curricula.

1.3 Hypothesis 1.3.1. H0: The effectiveness of DCM as educational tool is same to routine diabetic education among patients with diabetes type 2 (T2DM) visiting diabetic clinic in a tertiary care hospital of Karachi, Pakistan.

1.3.2. Ha: The effectiveness of DCM as educational tool is different to routine diabetic education among patients with diabetes type 2 (T2DM) visiting diabetic clinic in a tertiary care hospital of Karachi, Pakistan.

1.4 Objective of the study The objective of this study is to assess the effectiveness of DCM as an educational tool in comparison to routine care for improving the DMSE and DD among patients with type 2 diabetes mellitus visiting diabetic clinic of tertiary care hospital in Karachi, Pakistan.

1.5 Operational definitions

T2 Diabetes mellitus:

Type 2 diabetes is a metabolic condition where body develops resistance for insulin by progressive beta-cell dysfunction.

Diabetes control:

Patients with type 2 diabetes mellitus having HbA1c≤7

Diabetic Management Self-Efficacy (DMSE):

Patient level of confidence and believe that they can perform diabetes management activities such as, eat control diet, monitoring of blood glucose, administration of insulin/timely intake of oral medication , medical checkup, daily exercise in routine life in spite of challenging circumstances.

Suboptimal control of diabetes:

HbA1c is a clinical indicator, which shows how well diabetes is controlled for the last 3 months. HbA1c level more than 7 % will be considered suboptimal control of diabetes

Diabetes distress (DD):

Patient Experiences trouble and invisible emotional burdens, when managing a severe chronic disease like diabetes.

METHODOLOGY 1.1 Study Design: Randomized controlled trial 1.2 Study setting: This study will be conducted in National Institute of Diabetes and Endocrinology (NIDE) Ojha campus Dow University of Health Sciences (DUHS).

1.3 Study duration: Duration for the study will be one year after the final approval of synopsis. 1.4 Sample size A study from China (41) reported mean DDS score of control and intervention group at baseline as 32.77±14.57 and 26.08±9.92 respectively. After intervention the respective scores were 22.79±4.95 and 30.09±12.14. Using these estimates, 95% confidence interval and 80% power of the test, the computed sample size was 88, 44 in each group. After adding attrition rate, a total of 120 subjects i.e. 60 in control arm and 60 in intervention arm will be included in the study. Since there are two hospitals, 30 participants in each group will be included from each hospital.

1.5 Sampling technique Individual randomization will be done by opening the sealed envelopes for the allocation of intervention. There will be 120 sealed opaque envelopes containing either diabetes conversation map (acronym DCM; n=60) or routine care (acronym RC; n=60). These envelopes will be shuffled and opened for each eligible participant.

1.6 Data collection The principle investigator (PI) will take permission from related authority. The PI will be sitting in the waiting area outside the clinic where the physician will refer all the patients diagnosed with T2 diabetes with suboptimal management. After screening based on eligibility criteria, informed consent will be taken. Structured Questionnaire will be used for collecting demographic, clinical, and laboratory data.

After 3 months of enrollment, a follow up interview will be conducted using a structured questionnaire and blood test for HbA1c to see the change in baseline measurements across the two groups.

1.7 Intervention arm The intervention arm will receive 4 sessions based on diabetes conversation maps. These sessions will be conducted 1 week apart (45-60min) in a group of 5-8 participants per group. These sessions will be facilitated by a trained educator. These sessions will include topics on managing diabetes, following a healthy lifestyle, starting insulin, and experiencing life with diabetes.

Conversation Map (CM) education tools are a series of tools for facilitated group education 5-8 that were developed by Healthy Interactions in collaboration with the International Diabetes Federation (IDF) and are sponsored by Lilly Diabetes.

CM-based education guides people with diabetes through a process with the aim of helping them understand and internalize information about their disease and generate insightful conclusions, which may then result in improved self-management decisions and actions.

1.8 Control Arm In control group, participants will attend their routine regular appointments to health care professional and receive instruction provided as part of routine care during the study period.

1.9 Ethical concerns Approval for ethical consideration will be taken from Institutional Review Board of DUHS. Written inform Consent will be taken from all the participants including permission to access their medical records. No individual information of study participants and organization will be published as the data and results published will be in aggregate form for maintaining the confidentiality of the study participants and organization. All the information about the study participants will be kept in lock and key.

1.10 Study Variables:

Dependent variables:

Diabetes Management Self-Efficacy (DMSE) and Diabetes Distress (DD) and HbA1c are dependent variable in this study.

Independent variables:

This will include age, gender, BMI, education level, occupation, marital status, time since diabetes diagnosis, time since diabetes treatment, type of treatment for Diabetes e.g. Tablets, insulin etc. use of smart phones, use of internet and monthly income.

1.11 Statistical Analysis: All statistical analysis will be performed using SPSS version 20. Intention to treat and per protocol analysis will be performed. Descriptive statistics will be reported by computing frequencies and percentages for categorical variables and means, standard deviation and ranges (minimum and maximum) values for continuous variables. Outcome variables will be calculated by summing the scores of respective scales. Repeated Measures ANOVA will be used to measure difference in HbA1C, DMSE and DDS between intervention and control arm. Sensitivity analysis will be run to measure effect of any missing observations on outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients of both gendersage 30-60 years diagnosed with type 2 diabetes mellitusfor at least 5 years, presenting at the diabetes clinics of study setting and considered by health care professional to have a suboptimal management of their disease.
* Patient having HbA1c more than 7 will be included
* Patients who have not participated in any diabetic educational program before.
* Patients who will be found to be diabetes distressed as recommended in diabetes distress (DD) screening tool

Exclusion Criteria:

* Patients with major disabilities, diagnosed with mental health problems/ cognitive pattern not intact and those with major diabetes related complications.
* Patients residing outside of Karachi or intended to leave the city during the study duration will be excluded.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Diabetes Management Self-Efficacy (DMSE) at 3 months: | at baseline and after 3 months of enrollment
  The change in DMSE will be measured using validated DMSE scale. The scale has 20 items comprised of 4 domains; 1) nutrition specific and weight, 2) medical treatment, 3) physical exercise, 4) blood sugar. Each item is scored on 11 point likert scale (0=completely unable to 10=completely able). Possible score ranges from 0 to 200, with higher score representing higher self-efficacy.
Change from baseline Diabetes distress (DD) 3 months: | baseline and 3 months of enrollment
  The change in DD will be screened using validated DD scale. The scale has two parts; part 1 is consisting of two items asking about feelings of overburden due to demands of living with diabetes and feelings of failure with diabetes routine; the aim of part 1 is to screen for the presence of DD. Part 1 will be administered before the enrollment of the patient to screen for the presence of DD. If DD is present, part 2 will begin consisting of 17 items to score the extent of DD. Each item is scored on a likert scale ranging from 1 (not a problem) to 6 (a very serious problem). According to the instructions of DDS scoring sheet, total DDS will be measured with mean score while dividing the sum of all items by 17.The mean score of ≥3 will be the threshold for being distressed.

SECONDARY OUTCOMES:
Change from baseline HbA1C at 3 months: | baseline and 3 months after enorllment
  Change in HbA1c level will be measured at baseline and 3 months after enrollment to see mean difference in the two measurements

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Qasim, MSc, Principal Investigator — Dow University of Health Sciences, Ojha Campus
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qasim R, Masih S, Yousafzai MT, Shah H, Manan A, Shah Y, Yaqoob M, Razzaq A, Khan A, Rohilla ARK. Diabetes conversation map - a novel tool for diabetes management self-efficacy among type 2 diabetes patients in Pakistan: a randomized controlled trial. BMC Endocr Disord. 2020 Jun 16;20(1):88. doi: 10.1186/s12902-020-00572-x. PMID 32546240
- [Derived] Qasim R, Masih S, Hussain M, Ali A, Khan A, Shah Y, Shah H, Yousafzai MT. Effect of diabetic counseling based on conversation map as compared to routine counseling on diabetes management self-efficacy and diabetic distress among patients with diabetes in Pakistan: a randomized controlled trial (study protocol). BMC Public Health. 2019 Jul 8;19(1):907. doi: 10.1186/s12889-019-7266-3. PMID 31286927